CLINICAL TRIAL: NCT03261349
Title: A Pilot Phase II Study of New Direct-Acting Antiviral Agent, HARVONI® (Ledipasvir/Sofosbuvir), for the Treatment of Genotype 1 or 2 HCV-Associated Indolent B-Cell Non- Hodgkin's Lymphoma
Brief Title: Antiviral Agent HARVONI® for the Treatment of HCV-associated Indolent B-Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201612066MIPB
Record Dates: First submitted 2017-08-09; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Indolent Lymphoma
Keywords: Follicular lymphoma; MALT lymphoma; Waldenström's macroglobulinemia; Hepatitis C virus
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia; Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Intervention Model Description: New Direct-Acting Antiviral Agent, HARVONI® (ledipasvir/sofosbuvir)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Anti-HCV (Ledipasvir and sofosbuvir) (Experimental): Harvoni® (90 mg ledipasvir and 400 mg sofosbuvir) one tablet daily for 12 weeks
  Interventions: Drug: Ledipasvir and sofosbuvir

INTERVENTIONS:
Drug: Ledipasvir and sofosbuvir — To assess whether Harvoni® (ledipasvir and sofosbuvir) could eradicate HCV and lead to durable complete remission of these lymphomas.
  Other Names: HARVONI®

SUMMARY:
We and other investigators have revealed an association between Hepatitis C virus (HCV) seropositivity and an increased risk of developing marginal zone B-cell lymphoma (MZ), lymphoplasmacytic lymphoma (LPL, also known as Waldenström's macroglobulinemia), follicular lymphoma (FL), and diffuse large B-cell lymphoma (DLBCL). The sustained virologic response (SVR) to treatment with interferon or pegylated (Peg)IFN with ribavirin was closely associated with the regression of HCV-associated B-cell NHL (mainly MZL, and LPL).

Currently, the second-generation direct-acting antiviral agents (DAAs), such as sofosbuvir, have been shown to have a higher cure rate, less side effects, and a shorter duration of therapy for chronic HCV infection. After the approval of DAA for HCV therapy, several recent anecdotal case reports showed that indolent low-grade B-cell NHLs regressed after HCV clearance by DAAs. It is noted that the time to complete remission of these lymphomas was around 20 to 24 weeks after starting DAAs. These findings indicate that DAAs can eradicate the trigger of lymphomagenesis by curing chronic HCV infection.

Because DAAs are more potent and efficient than pegylated (Peg) interferon plus ribavirin and well-tolerated for the treatment of HCV infection, it is reasonable to use DAAs as the frontline treatment for HCV-positive patients with indolent B-cell NHL, such as MZL, LPL, and low-grade FL, who do not require immediate cytoreductive therapy. The aim of this proposal is to assess whether Harvoni® (ledipasvir and sofosbuvir) could eradicate HCV and lead to durable complete remission of these lymphomas..

DETAILED DESCRIPTION:
Although several epidemiological studies, including our study have been demonstrated the link between HCV and B-cell non-Hodgkin's lymphoma (NHL), the direct evidence of the HCV-associated-NHL remains uncertain. Direct antiviral agents (DAA) have been shown to have a higher cure rate, less side effects, and a shorter duration of therapy for chronic HCV infection. Whether DAA treatment can cure HCV-associated indolent B-cell NHL remains unclear? If yes, a direct evidence of HCV-associated lymphomagenesis will be approved. Because DAAs are more potent and efficient than pegylated (Peg) interferon plus ribavirin and well-tolerated for the treatment of HCV infection, it is reasonable to use DAAs as the frontline treatment for HCV-positive patients with indolent B-cell NHL, such as MZL, LPL, and low-grade FL, who do not require immediate cytoreductive therapy. The aim of this proposal is to assess whether Harvoni® (ledipasvir and sofosbuvir) could eradicate HCV and lead to durable complete remission of HCV-associated indolent B-cell NHL.

In the translational part, we will assess the expression pattern of BAFF-related canonical and non-canonical NF-κB signaling molecules by immunohistochemical (IHC) staining, and t(11;18)(q21;q21), and t(14;18)(q32;q21) by fluorescence in situ hybridization (FISH) in pre-treatment tumors samples of patients in prospectively predicting the antiviral responsiveness of HCV-positive indolent B-cell NHLs. The serum cytokines and chemokines, IFN-gamma, TNF-alpha, IL-4, IL-5, IL-6, IL-13 and CXCL13, BAFF level, and HCV RNA load before and after DAA treatment in HCV-associated indolent B-cell NHLs will be examined. The genotype of the HLA class II, and cloning followed by sequences of the VH region of the immunoglobulin gene derived from pre-treatment tumor samples will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years with histologically proven diagnoses of indolent B-cell NHLs and with positive genotype 1 or 2 HCV (non-cirrhotic status) were eligible.
2. Indolent B-cell NHLs includes:

   * Low-grade marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue (MALT) type: known as MALT lymphoma.
   * Splenic marginal zone lymphomas (SMZL)
   * Waldenström's macroglobulinemia (WM, known as lymphoplasmacytic lymphoma) .
   * Grade 1, 2 follicular lymphoma (FL). 3 Stage I to III (modified Ann Arbor stage), and non-life threatening IV lymphoma. 4 Patients had not previously been treated with chemotherapy or immunotherapy, were eligible. 5 Patients with clinical, echographical, or radiological suspicion of lymphoma lesions were eligible.

Exclusion Criteria:

1. Evidence of histologic transformation to a high-grade lymphoma (such as grade 3 and 4 follicular lymphoma, and high-grade MALT lymphoma).
2. Life-threatening disseminated lymphoma.
3. Primary gastric lesions were not eligible.
4. Prior diagnosis of neoplasm within 5 years, except cervical intraepithelial neoplasia type 1 (CIN1) or localized non-melanomatous skin cancer.
5. Evidence of clinically significant cardiac disease, as defined by history of symptomatic ventricular arrhythmias, congestive heart failure or myocardial infarction within 12 months before study entry.
6. Evidence of symptomatic central nervous system (CNS) disease.
7. Evidence of active opportunistic infections.
8. Liver cirrhosis B and C (Child-Pugh score)
9. Known HIV infection.
10. Pregnant or lactating status.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-08-15 (Estimated)

PRIMARY OUTCOMES:
The complete remission rate | During the first-year, every 3 months to evaluate
  The complete remission rate by using Harvoni® (ledipasvir and sofosbuvir) as the first-line line therapy.

SECONDARY OUTCOMES:
The durability of complete remission (disease-free interval) | Follow-up every 3 motnhs for 3 years
  The lymphoma-free
The overall response rate | During the first-year, every 3 months to evaluate
  Complete remission and partial remission rate
The association between HCV RNA load and response of lymphoma. | During the first-year, every 3 months to evaluate
  The assessment of HCV RNA load
The toxicity of Harvoni®. | 3 months
  The assessment of toxicity during the first 3 months
Potential biomarkers predicting the response of Harvoni®. | 3 years
  Translational study

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Hsin Kuo, M.D.,Ph.D., Principal Investigator — Department of Oncology, National Taiwan University Hospital